CLINICAL TRIAL: NCT04747171
Title: A Comparative Study of Postoperative Analgesia of Different Intrathecal Additives for Spinal Anaesthesia in Elective Caesarean Sections
Brief Title: Intrathecal Additives for Spinal Anaesthesia in Elective Caesarean Sections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Baher Said Elshahat Mohamed Abdelhady, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: spinal additives
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- magnesium intrathecal (Active Comparator)
  Interventions: Drug: intrathecal Magnesium
- dexamethasone intrathecal (Active Comparator)
  Interventions: Drug: intrathecal dexamthasone
- dexmedetomidine intrathecal (Active Comparator)
  Interventions: Drug: intrathecal dexmedetomidine

INTERVENTIONS:
Drug: intrathecal Magnesium — intrathecal adjuvants to bupivacaine
  Arms: magnesium intrathecal
Drug: intrathecal dexamthasone — intrathecal adjuvants to bupivacaine
  Arms: dexamethasone intrathecal
Drug: intrathecal dexmedetomidine — intrathecal adjuvants to bupivacaine
  Arms: dexmedetomidine intrathecal

SUMMARY:
we designed this randomized, single -blind, prospective clinical study to test postoperative analgesia of three intrathecal additives in elective caesarean sections which are magnesium, dexamethasone and dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classII-III adult female patient (age :18 -40 years old )
* Elective cesarean section under spinal anaesthesia
* Gestational age > 37 weeks
* BMI less than 30 kg/m2

Exclusion Criteria:

* Patient refusal
* unable to give consent
* age < 18 or > 40
* BMI more than 30 kg/m2
* known allergy to the study medication
* coagulopathies or on anticoagulant medications
* diabetic neuropathy
* patients with psychiatric disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
analgesic effect | Up to 24 hours after surgery
  duration of sensory block